CLINICAL TRIAL: NCT01833312
Title: EuroHYP-1: European Multicentre, Randomised, Phase III Clinical Trial of Therapeutic Hypothermia Plus Best Medical Treatment Versus Best Medical Treatment Alone for Acute Ischaemic Stroke
Brief Title: Cooling Plus Best Medical Treatment Versus Best Medical Treatment Alone for Acute Ischaemic Stroke
Acronym: EuroHYP-1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow recruitment, cessation of funding
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EuroHYP-1
Record Dates: First submitted 2013-04-04; First posted 2013-04-16 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stroke; hypothermia
MeSH Terms: conditions — Ischemic Stroke; Hypothermia | interventions — Buspirone; Meperidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypothermia (Experimental): Best medical treatment + hypothermia 34-35°C for 24h
  Interventions: Device: Hypothermia; Drug: Buspirone; Drug: Pethidine
- Control (No Intervention): Best medical treatment

INTERVENTIONS:
Device: Hypothermia — In patients randomised to therapeutic hypothermia, induction of cooling will be started by infusion of 4°C isotone saline or Ringer's lactate administered over a period of 30 to 60 minutes. A body temperature between 34.0 and 35.0°C will be targeted. Body temperature will be monitored through bladder or rectal thermal probes, and cooling procedures will be adapted to keep body temperature as close as possible to the target. Maintenance of body temperature in the target range will be performed with a surface or endovascular cooling device. After a cooling period of 24h, controlled rewarming to 36°C with a rate of 0.2°C/h will be started. After 36°C have been reached, the device will be disconnected.
  Other Names: EMCOOLS Brain.Pad; Arctic Sun and ArcticGel Pads; CritiCool and CureWrap 3500; Zoll intravascular temperature management system
  Arms: Hypothermia
Drug: Buspirone — anti-shivering treatment
  Arms: Hypothermia
Drug: Pethidine — anti-shivering treatment
  Arms: Hypothermia

SUMMARY:
The purpose of this study is to determine if systemic cooling to a target temperature of 34 to 35°C, started within 6 hours of symptom onset and maintained for 12 hours, improves functional outcome at 3 months in patients with acute ischaemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the patient or his/her legally acceptable representative or under such other arrangements as may be legally established in participating countries
* Patients of both sexes aged ≥18 years
* Estimated body weight of 50 up to and including 120kg
* Diagnosis of acute ischaemic stroke
* Possibility to start therapeutic hypothermia within 6 hours after onset of stroke
* Possibility to start therapeutic hypothermia within 150 minutes after start of alteplase administration in patients receiving thrombolysis at the trial site or within 150 minutes after start of endovascular treatment, if this is later
* Possibility to start therapeutic hypothermia within 150 minutes after admission to trial site in patients not receiving thrombolysis or in patients who have received thrombolysis at a different site
* mRS score ≤2 prior to onset of stroke
* NIHSS score ≥6
* GCS motor response subscale score ≥5

Exclusion Criteria:

* Use of monoamineoxidase inhibitors in the 14 days prior to screening
* Current use of medication interacting with pethidine or buspirone, i.e., ritonavir, phenytoin, cimetidine, phenothiazines, opioids and partial opioid agonists (e.g., pentazocine, nalbuphine, buprenorphine)
* Acute alcohol intoxication
* Opioid addiction
* Nursing mother or pregnant woman, as verified by a positive urine pregnancy test in females of childbearing potential
* Known hypersensitivity to the IMPs or any of their formulation ingredients
* Patient who is imprisoned or is lawfully kept in an institution
* Employee or direct relative of an employee of the CRO (if applicable), the department of the investigator, or the sponsor
* Participation in an interventional clinical trial within the last 4 weeks, or be under the exclusion period from another trial
* Prior participation in this trial
* Any acutely life-threatening conditions other than acute ischaemic stroke
* Rapidly resolving stroke symptoms
* Evidence from CT or MRI of intracranial haemorrhage or tumour or encephalitis or any diagnosis likely to cause the present symptoms other than acute ischaemic stroke. Haemorrhagic transformation of the infarct is not an exclusion criterion, except when there is a parenchymal haematoma covering more than 30% of the infarcted area, with significant space-occupying effect, or when there is a bleeding remote from the infarcted area
* Known convulsive disorder, acute closed angle glaucoma, myasthenia gravis
* SPO2 <94% (as measured by pulse oximetry) under nasal oxygen administration
* Other severe respiratory disorder
* Bradycardia (<40 bpm)
* Severe cardiac failure, defined as NYHA classification ≥III
* Myocardial infarction or angina pectoris in the 3 months prior to screening
* Vasospastic disorders (e.g., Raynaud's disease)
* Haematological dyscrasia (e.g., sickle cell disease, cryoglobulinaemia)
* Known platelet count <100,000/mm3
* Known INR >1.7
* Skin damage (e.g., inflammation, burns, injuries, ulcerations, hives, rash) at the sites intended to be used for cooling
* Clinical diagnosis of sepsis
* Known severe hepatic impairment (serum ALAT and/or ASAT >3 times ULN)
* Known renal impairment (serum creatinine >2mg/100ml)
* Addison's disease
* Any other condition that may interfere with, or be aggravated by, therapeutic hypothermia
* Any condition that is thought to reduce the compliance to cooperate with the trial procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2013-07; Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
modified Rankin scale | 3 months
  Analysed with ordinal logistic regression and expressed as a common odds ratio.

SECONDARY OUTCOMES:
Mortality | 3 months
Neurological outcome | 3 months
  NIHSS;
  World Health Organization Disability Assessment Schedule (WHODAS) 2.0
Quality of life | 3 months
  EuroQoL 5-dimensions 5-level questionnaire
Cerebral infarct size | 48±24 hours
  Evaluated on CT or MRI imaging
Safety of systemic cooling | Enrollment - day 91
  Number of adverse events and severe adverse events related to the procedure of systemic cooling including induction, maintenance of hypothermia, rewarming, or the administration of anti-shivering medication (pethidine and buspirone) within the first 36h of enrollment.
  Number of adverse events and severe adverse events until outcome assessment at day 91.
Tolerability of systemic cooling | 36 hours
  Timing and dose of anti-shivering medication.
  Bedside shivering assessment scale (BSAS).

OTHER OUTCOMES:
Selected biomarkers | baseline, 24h, 72h
  * MMPs including gelatinases (MMP-2 and MMP-9), collagenases (MMP-1, MMP-8 and MMP-13) and stromelysins (MMP-3 and MMP-10) using multiplex ELISA [SearchLight technology].
  * MMP endogen inhibitors (TIMP-1 and TIMP-2) using multiplex ELISA [SearchLight technology].
  * H-FABP, UFD-1, RNABP, NDKA, GSTP-1 and Pro-BNP using standard ELISA.
  * Cerebral Array I & II containing BDNF, GFAP, NSE, NGAL, sTNFRI, D-dimer and CRP using biochip analysers [Randox].
  * Pro-ANP, Copeptin, IL6, IL8, IL10, mannose-binding lectin (MBL), mHLA-DR, monocytotic cytokine-secretion ex vivo stimulation, C5a in plasma, ultrasensitive PCT, lipopolysaccharide-binding protein (LBP).
Other imaging parameters | baseline, 48h
  Presence, location and extent of any visible infarct, early infarct swelling, hyperdense artery, leukoaraiosis, atrophy and prior infarct on the scan performed at screening assessment (within 90 minutes before the start of the treatment) will be tested for any interaction with early (infarct swelling, haemorrhagic transformation, neurological deterioration, death) and late (NIHSS and mRS scores, death) neurological and functional outcome variables at day 8 or day of discharge from hospital, whichever occurs firs, and at outcome assessment (day 91±14).
Cost-effectiveness parameters | 3 months
  Patient location during stay in hospital.
  Destination after discharge from hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Schwab, Prof, Study Chair — University of Erlangen-Nürnberg
Locations (1):
- Department of Neurology, University Hospital Erlangen, Erlangen, Germany

REFERENCES:
- [Derived] Winkel P, Bath PM, Gluud C, Lindschou J, van der Worp HB, Macleod MR, Szabo I, Durand-Zaleski I, Schwab S; EuroHYP-1 trial investigators. Statistical analysis plan for the EuroHYP-1 trial: European multicentre, randomised, phase III clinical trial of the therapeutic hypothermia plus best medical treatment versus best medical treatment alone for acute ischaemic stroke. Trials. 2017 Nov 29;18(1):573. doi: 10.1186/s13063-017-2302-z. PMID 29187242
- [Derived] van der Worp HB, Macleod MR, Bath PM, Demotes J, Durand-Zaleski I, Gebhardt B, Gluud C, Kollmar R, Krieger DW, Lees KR, Molina C, Montaner J, Roine RO, Petersson J, Staykov D, Szabo I, Wardlaw JM, Schwab S; EuroHYP-1 investigators. EuroHYP-1: European multicenter, randomized, phase III clinical trial of therapeutic hypothermia plus best medical treatment vs. best medical treatment alone for acute ischemic stroke. Int J Stroke. 2014 Jul;9(5):642-5. doi: 10.1111/ijs.12294. Epub 2014 May 15. PMID 24828363